CLINICAL TRIAL: NCT06068790
Title: 28Fr Versus 22Fr HoLEP, a Randomized Controlled Trial Indiana University School of Medicine, Department of Urology
Brief Title: Incontinence Analysis After HoLEP Using 28Fr Versus 22Fr Sheath
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No Current scope was available to perform procedure.
Sponsor: Marcelino Rivera (Other)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor-Investigator, Marcelino Rivera, Assistant Professor of Urology, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IndianaU 14563
Record Dates: First submitted 2023-08-29; First posted 2023-10-05 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: We hypothesize there will be lower rates of immediate urinary incontinence, and urethral stricture formation in patients undergoing HoLEP with smaller 22Fr sheaths compared to 28 Fr.
Masking Description: This study will be a randomized controlled trial in which patients who meet inclusion criteria will be randomized to one of two groups, HoLEP performed with either 1) 22Fr sheath set or 2) 28Fr sheath set. After HoLEP, data will be analyzed using chi-square test for incontinence vs no incontinence between 22Fr and 28Fr groups at 1 week, 4 weeks and 12 weeks post operatively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HoLEP surgery with 22Fr (Active Comparator): HoLEP will be performed per standard clinical care with the instruments assigned at randomization - 22Fr or 28Fr.
  Interventions: Device: 22 French sized rigid sheath
- HoLEP surgery with 28Fr (Experimental): HoLEP will be performed per standard clinical care with the instruments assigned at randomization - 22Fr or 28Fr.
  Interventions: Device: 28 French sized rigid sheath

INTERVENTIONS:
Procedure: HoLEP Surgery — HoLEP will be performed per standard clinical care with the instruments assigned at randomization - 22Fr or 28Fr.
Device: 28 French sized rigid sheath — The 28Fr is the standard of care sheath size used at this site.
  Other Names: 28Fr
  Arms: HoLEP surgery with 28Fr
Device: 22 French sized rigid sheath — The 22Fr is the smaller, investigational sheath size to be used in this study.
  Other Names: 22Fr
  Arms: HoLEP surgery with 22Fr

SUMMARY:
The rationale for this study is to assess whether there is a difference in HoLEP outcomes in smaller 22Fr instruments compared to our standard 28Fr sheaths.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial in which patients who meet inclusion criteria will be randomized to one of two groups, HoLEP performed with either 1) 22Fr sheath set or 2) 28Fr sheath set. After HoLEP, data will be analyzed using chi-square test for incontinence vs no incontinence between 22Fr and 28Fr groups at 1 week, 4 weeks and 12 weeks post operatively.

ELIGIBILITY:
Inclusion Criteria:• Age >18 years old Undergoing HoLEP for benign prostatic enlargement Eligible for same day catheter removal

Exclusion Criteria:

* Age < 18 years old
* Existing stress or urge urinary incontinence
* Planned overnight admission or overnight catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Assessing differences in HoLEP outcomes in smaller 22Fr instruments compared to our standard 28Fr sheaths. | M-ISI survey completed at 1,4,12 weeks
  Measuring rates of immediate urinary incontinence or complications post-operation HoLEP using the Michigan Incontinence System Index (M-ISI) survey.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Indiana University Health Physicians Urology, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana